CLINICAL TRIAL: NCT06888453
Title: Evaluation the Effects of Propolis Lozenges Extract on Salivary Biomarkers and Its Effect on Oral Health Condition in (19_24) Years Old
Brief Title: Propolis Lozenges Extract and Their Effect on Salivary Biomarkers and on Oral Health Condition in (19_24) Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Ahmed Salah Abdulmahdi Finajn, master student, Al-Mustansiriyah University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL-Mustansiriyah University
Record Dates: First submitted 2025-03-05; First posted 2025-03-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Plaque Induced Gingivitis; Mouth Diseases; Periodontal Diseases
Keywords: gingivitis; plaque; propolis; lozenges
MeSH Terms: conditions — Mouth Diseases; Periodontal Diseases; Gingivitis; Plaque, Amyloid | interventions — Propolis

STUDY DESIGN:
Intervention Model Description: 100 subjects with plaque induced gingivitis, caused by accumulation of plaque, will be selected and enrolled in this study. Subsequently, subjects will be equally divided case and control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lozenges containing propolis (Experimental): lozenges containing propolis Participants will be given the test interventions, lozenges containing propolis, and will be asked to chew twice per day and will be instructed to ordinary oral hygiene instruction, No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.
  Interventions: Drug: lozenges containing propolis
- standard of care (No Intervention): Participants will be instructed to ordinary oral hygiene instruction only, No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days.

INTERVENTIONS:
Drug: lozenges containing propolis — lozenges containing propolis Participants will be given the test interventions, lozenges containing propolis, and will be asked to chew twice per day and will be instructed to ordinary oral hygiene instruction, No modifications to the participants' tooth brushing technique will be permitted. Next, the participants will be re-evaluated after 7 days
  Other Names: bee glue
  Arms: lozenges containing propolis

SUMMARY:
The goal of this clinical trial is to test the efficiency of using lozenges containing propolis extract over one week to control gingival inflammation and plaque accumulation by measuring the clinical periodontal parameters (Gingival index, plaque index) in comparison with a control group given oral hygiene instruction only in patients with biofilm induced gingivitis (moderate gingivitis)

Objectives:

1. Evaluate the clinical efficiency of using lozenges containing propolis extract over 7 days to control gingival inflammation and plaque accumulation by measuring the clinical periodontal parameters (Gingival index, plaque index) in comparison with a control group given oral hygiene instruction only in patients with biofilm induced gingivitis (moderate gingivitis).
2. Measuring levels of salivary cytokines, IL-1Beta, and IL-10 by ELISA at Baseline visit before using lozenges containing propolis and after 7 days of using lozenges containing propolis compared to a control group with oral hygiene instruction only.
3. Investigate and compare the association of salivary interleukins of IL-Beta and IL-10 in periodontal health and generalized gingivitis.
4. Evaluate the correlation between clinical periodontal parameters and salivary (IL-1Beta and IL-10).
5. Evaluate subjects' perception of lozenges containing propolis extract and oral hygiene instructions after 7 days.

DETAILED DESCRIPTION:
100 subjects will be enrolled, who show generalized gingivitis (moderate gingivitis) with no Periodontal pocket depth>3 mm, intact periodontium, and no loss of periodontal attachment), caused by the accumulation of plaque. 50 subjects are case that given a lozenge containing propolis and oral hygiene instructions, and 50 subjects were control that were given oral hygiene instructions only. The participants will be asked to chew a lozenge twice per day and Discontinuation of the lozenges will be advised in cases of any allergic reaction. in baseline visit at the beginning, Saliva collection for IL-1β and IL-10 measurement, then clinical periodontal parameters examination starting with gingival index (Loe and Silness in 1963) designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency, and bleeding on probing. A periodontal probe will be run along the gingival margin. The gingiva surrounding the tooth is assessed at four sites: mesio-facial papilla, facial marginal gingiva, disto-facial papilla and lingual marginal gingiva. Then finally followed by the Plaque Index (Loe and Silness in 1963). the data had been recorded from labial/buccal and lingual/palatal surfaces.

First visit after 7 days, from the baseline visit. Saliva collection and clinical periodontal parameters scoring (GI, PI) will be performed again as described at the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age of patients (19_24) who volunteered to participate.
2. Apparently, good general health. With no systemic diseases.
3. plaque and gingival indices were ranged from (1.1_2.0)

Exclusion Criteria:

* 1. Individuals with chronic illnesses, immunocompromised individuals, pregnant women, those on contraceptive medications, and breastfeeding mothers.

  2. People who use mouthwash at the moment or any preventive modalities. 3. Those taking anti-inflammatory drugs and antibiotics both during the study and in the final four weeks prior.

  4. Individuals have a history of hypersensitivity to any substance utilized in the current investigation.

  5. Individuals who have undergone a recent tooth extraction. 6. Individuals with Periodontal pocket depth Equal or less than 4 or attachment loss.

  7. Individuals who smoke. 8. Individuals with orthodontic equipment, removable dentures, implants.

Ages: 19 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2025-03-23 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Changes in the clinical periodontal parameter (Gingival index) | (0, 7days)
  Subjects will undergo the measurement of the gingival index according to (Loe & Silness in 1963), designed to assess the severity and quality of gingival inflammation in an individual or population. The gingival inflammation is assessed on the basis of color, consistency, and bleeding on probing. The Gingival Index (GI) scores each site on a 0 to 3 scale
  Score 0 : Normal gingiva
  score 1: Mild Inflammation- slight change in color, Slight oedema. No bleeding on probing.
  score 2: Moderate inflammation-redness, oedema and glazing. Bleeding on probing.
  score 3: Sever inflammation-marked redness and edema. Ulceration. Tendency to spontaneous bleeding.

SECONDARY OUTCOMES:
Changes in the clinical periodontal parameter (Plaque index ) | (0, 7days)
  To determine the patients' plaque index, their dental plaque thickness was evaluated by probing the mesial, distal, buccal, and palatal surfaces of all teeth using a Williams periodontal probe. The individual's plaque index was determined by summing the values obtained for each tooth and calculating the averages.Silness & Löe (Silness & Löe,1964) reference values were taken as a basis The Plaque Index (PI) scores each site on a 0 to 3 scale
  Score 0 : No plaque is in the area adjacent to the gingiva.
  Score 1: There is a plaque in the form of a thin film on the gingival margin.
  Score 2: There is a visible plaque in the gingival pocket and gingival margin.
  Score 3: There is a dense plaque in the gingival pocket and on the gingival margin.
Changes in salivary cytokines (IL- 1β , IL-10) | (0, 7days)
  ELISA kit will analyze salivary interleukins, and concentrations are measured according to manufacturing instructions, were picogram per liter for interleukin 1 beta levels and nanogram per milliliter for interleukin 10 levels
  0 day: Saliva collection for IL-1β and IL-10 measurement, then clinical periodontal parameters examination starting with the gingival index finally followed by the Plaque index
  7 days: Saliva collection and clinical periodontal parameters scoring (GI, PI) will be performed again as described at the baseline visit,

CONTACTS AND LOCATIONS:
Overall Officials: ahmed s aljanaby, B.D.S, Principal Investigator — Al-Mustansiriyah University; mohammed K Mahmoud, M.S.C, Study Director — Al-Mustansiriyah University
Locations (1):
- Almustansiriyah University, Baghdad, Iraq

REFERENCES:
- [Background] Shi H, Yang H, Zhang X, Yu LL. Identification and quantification of phytochemical composition and anti-inflammatory and radical scavenging properties of methanolic extracts of Chinese propolis. J Agric Food Chem. 2012 Dec 19;60(50):12403-10. doi: 10.1021/jf3042775. Epub 2012 Dec 5. PMID 23176258
- [Background] El-Allaky HS, Wahba NA, Talaat DM, Zakaria AS. Antimicrobial Effect of Propolis Administered through Two Different Vehicles in High Caries Risk Children: A Randomized Clinical Trial. J Clin Pediatr Dent. 2020 Sep 1;44(5):289-295. doi: 10.17796/1053-4625-44.5.1. PMID 33181849
- [Background] Alghutaimel H, Matoug-Elwerfelli M, Alhaji M, Albawardi F, Nagendrababu V, Dummer PMH. Propolis Use in Dentistry: A Narrative Review of Its Preventive and Therapeutic Applications. Int Dent J. 2024 Jun;74(3):365-386. doi: 10.1016/j.identj.2024.01.018. Epub 2024 Feb 19. PMID 38378400

DOCUMENTS (1):
  • Informed Consent Form (2024-11-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT06888453/ICF_000.pdf